CLINICAL TRIAL: NCT02269020
Title: Unilateral Selective Neck Dissection at Lymph Node Levels IIa, III and IV Using a Robot-assisted Transaxillary Approach in Patients With Squamous Cell Carcinoma of the Epi-larynx: the First Three Patients
Brief Title: Neck Dissection Via a Robot-assisted Transaxillary Approach in Patients With Squamous Cell Carcinoma of the Epi-larynx
Acronym: RoboCurage ORL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2013/BL-01; 2014-A00117-40 (Other: RCB number)
Record Dates: First submitted 2014-10-08; First posted 2014-10-20 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Squamous Cell Carcinoma of the Epi-larynx
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Neck Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3 patients cancer of the epi larynx (Experimental): 3 patients with squamous cell carcinoma of the epi-larynx
  Intervention: Neck Dissection
  Interventions: Procedure: Neck Dissection

INTERVENTIONS:
Procedure: Neck Dissection — Unilateral Selective Neck Dissection at Lymph Node Levels IIa, III and IV Using a Robot-assisted Transaxillary Approach. The robotic system used is the da Vinci system.

SUMMARY:
The main hypothesis of this study is that it is possible to make a unilateral selective dissection of ganglion levels IIa, III and IV using an endoscopic transaxillary approach via the da Vinci robotic system to reduce scarring, while respecting patient safety.

Feasibility will be assessed by two combinded criteria: 1) performance of the surgical procedure respecting the different stages of visualization and dissection of key anatomical elements; 2) obtain a minimum of 9 lymph nodes when analyzing pathological evidence of the dissection.

DETAILED DESCRIPTION:
Secondary objectives include the following:

A. Describe certain technical variables: surgical time, extent of blood loss, need for conversion to open surgery, anesthesia procedure used, the level of difficulty and speed associated with each surgical step, length of stay, B. Describe the pathological findings for each patient, C. Evaluate neurological complications (function of cranial nerve pairs X, XI, XII, brachial plexus, cervical sympathetic) D. Identify specific complications, E. Evaluate post-operative pain, F. Evaluate the scar outcome at 6 and 12 months G. Describe the oncological results at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the epi-larynx: (i) ranked T1 or T2 in the TNM classification, (ii) supraglottic or glotto-supraglottic location, (iii) CN0 nodal status
* Absence of distant metastasis (M0)
* Decision for unilateral endoscopic axillary neck dissection at lymph node levels IIa, III and IV of the Robins classification is retained in a multidisciplinary meeting
* The patient is available for 12 months of follow-up
* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan

Exclusion Criteria:

* Patient participating in or having participated in another study within the previous 3 months or currently in an exclusion period determined by a previous study
* Adult under judicial protection or any kind of guardianship
* Refusal to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Preoperative diagnosis of a second location of cancerous disease
* Body Mass Index > 25
* History of cervical spine surgery
* History of instability of the cervical spine
* History of surgery in the shoulder or pre-pectoral region
* History of ipsilateral neck surgery
* History of cervical radiotherapy
* History of breast implants

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Number of patients that had pre-defined key points of the surgical procedure performed | Day 0
  Were all pre-defined key points of the surgical procedure performed? yes/no Description of the key points (includes (i) axillary approach, (ii) robot arm insertion, (iii) dissection, (iv) closing) of the surgical procedure.
Number of lymph nodes dissected | Day 0
  Determined by analysis of excised tissues.

SECONDARY OUTCOMES:
The duration of surgical site preparation | Day 0
  in minutes
The duration of robot installation / preparation | Day O
  in minutes
Intervention time (between incision and closure by the surgeon) | Day 0
  in minutes
Time in general anesthesia | Day 0
  in minutes
Surgical time (console time for robot-assisted surgery) | Day 0
  in minutes
The estimated volume of bleeding | Day 0
  in ml
Need for conversion to open surgery | Day 0
  yes/no
The anesthesia protocol used | Day 0
  Full description.
The level of difficulty associated with each surgical step | Day 0
  Qualitative: easy, medium, hard, extremely hard
The level of speed associated with each surgical step | Day 0
  Qualitative: slow, normal, fast
Length of hospital stay in days | estimated max of 6 days
Results of pathological analysis of lymph nodes | expected between day 7 and day 15

OTHER OUTCOMES:
The number of ganglions excised at each level. | expected between day 7 and day 15
The number of metastatic ganglions | expected between day 7 and day 15
The presence/absence of capsular rupture | expected between day 7 and day 15
Normal functioning of cranial nerve IX: yes/no. | Day 15
Normal functioning of cranial nerve X: yes/no. | Day 15
Normal functioning of cranial nerve XI: yes/no. | Day 15
Normal functioning of cranial nerve XII: yes/no. | Day 15
Normal functioning of the brachial plexus nerve: yes/no. | Day 15
Normal functioning of the cervical sympathetic nerve: yes/no. | Day 15
Normal functioning of cranial nerve IX: yes/no. | Month 6
Normal functioning of cranial nerve X: yes/no. | Month 6
Normal functioning of cranial nerve XI: yes/no. | Month 6
Normal functioning of cranial nerve XII: yes/no. | Month 6
Normal functioning of the brachial plexus nerve: yes/no. | Month 6
Normal functioning of the cervial sympathetic nerve: yes/no. | Month 6
Normal functioning of cranial nerve IX: yes/no. | Month 12
Normal functioning of cranial nerve X: yes/no. | Month 12
Normal functioning of cranial nerve XI: yes/no. | Month 12
Normal functioning of cranial nerve XII: yes/no. | Month 12
Normal functioning of the brachial plexus nerve: yes/no. | Month 12
Normal functioning of the cervical sympathetic nerve: yes/no. | Month 12
Presence/absence of intraoperative complications | Day 0
Presence / absence of complications during the hospitalization period | estimated max of 6 days
Presence / absence of complications at the post-operative follow-up visit | day 7 to day 15
Analgesic consumption | During hospitalization; expected max of 6 days
  Qualitative: Level I, Level II, Level III.
Analgesic consumption | days 7 to 15
  Qualitative: Level I, Level II, Level III.
Analgesic consumption | month 6
  Qualitative: Level I, Level II, Level III.
Daily visual analog scale for pain | During hospitalization; expected max of 6 days.
Visual analog scale for pain | days 7 to 15
Visual analog scale for pain | month 6
Visual analog scale for pain | month 12
Length of axillary scar | day 0
Length of thoracic scar | day 0
Length of axillary scar | month 6
Length of thoracic scar | month 6
Length of axillary scar | month 12
Length of thoracic scar | month 12
Patient satisfaction concerning his/her scar | month 6
  visual analog scale from 0 to 10
Patient satisfaction concerning his/her scar | month 12
  visual analog scale from 0 to 10
Oncological results | month 6
  Qualitative variable: (A) Living with disease progression, if so: (i) Recurrence: yes / no; (ii) Metastases: yes / no. or (B) Living without recurrence or (C) Deceased; give causes.
Oncological results | month 12
  Qualitative variable: (A) Living with disease progression, if so: (i) Recurrence: yes / no; (ii) Metastases: yes / no. or (B) Living without recurrence or (C) Deceased; give causes.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lallemant, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France